CLINICAL TRIAL: NCT05226819
Title: Analysis of Influencing Factors of Helicobacter Pylori Infection and Eradication Failure in Outpatients of Digestive Department in Xi'an
Brief Title: Influencing Factors of Helicobacter Pylori Infection and Eradication Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020065
Record Dates: First submitted 2022-01-08; First posted 2022-02-07 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Infection; Risk Factor; Questionnaire
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- H. pylori negative group (No Intervention): No Intervention
- H. pylori positive and successful eradication group (Other): H. pylori-positive patients are given rabeprazole 10mg + amoxicillin 1000mg + clarithromycin 500mg + colloidal bismuth tartrate 220mg bid for 14 days. After 4-6 weeks of completing eradication therapy, 13C-UBT is performed and the result show that H. pylori is eradicated. At the same time, Patients with successful eradication are instructed to conduct 13C-UBT examination after 6 months,1year and every year after drug withdrawal.
  Interventions: Drug: PPI quadruple therapy
- H. pylori positive and eradication failure group (Other): H. pylori-positive patients are given rabeprazole 10mg + amoxicillin 1000mg + clarithromycin 500mg + colloidal bismuth tartrate 220mg bid for 14 days. After 4-6 weeks of completing eradication therapy, 13C-UBT is performed and the result show that H. pylori is not eradicated.
  Interventions: Drug: PPI quadruple therapy

INTERVENTIONS:
Drug: PPI quadruple therapy — Among these outpatients, H. pylori-negative patients don't give any intervention. But H. pylori-positive patients are given rabeprazole 10mg + amoxicillin 1000mg + clarithromycin 500mg + colloidal bismuth tartrate 220mg bid for 14 days. After 4-6 weeks of completing eradication therapy, 13C-UBT is performed.
  Arms: H. pylori positive and eradication failure group; H. pylori positive and successful eradication group

SUMMARY:
Helicobacter pylori (H. pylori) is closely related to the occurrence of gastric cancer and other diseases, the discovery and eradication of H. pylori infection has great significance to the prevention and treatment of related diseases. At the same time,understanding the influencing factors of H. pylori infection and eradication failure in the population can provide a scientific basis for the formulation of local H. pylori prevention and control strategies. So, the investigators intend to analyze the factors related to H. pylori infection and eradication failure in the outpatients of gastroenterology clinics in Xi'an, China.

DETAILED DESCRIPTION:
Taking 300 permanent residents in Xi'an area who will go to the Gastroenterology Clinic of the Second Affiliated Hospital of Xi'an Jiaotong University from February 2022 to March 2023 and undergo 13C-UBT examination as the research object. A questionnaire survey on factors related to H. pylori infection and eradication failure will be conducted. The questionnaire includes basic Information, eating patterns, living environment, related gastrointestinal symptoms, etc. Among the outpatients, H. pylori-positive patients will be given rabeprazole 10 mg + amoxicillin 1000 mg + clarithromycin 500 mg + colloidal bismuth tartrate 220 mg bid for 14 days. After 4-6 weeks of completing eradication therapy, 13C-UBT will be performed to determine whether H. pylori is eradicated. According to the results of 13C-UBT at the beginning and results of 13C-UBT after eradication treatment, outpatients will be divided into three groups: H. pylori negative group, H. pylori positive radical cure successful group and H. pylori positive radical cure failed group. Next using SPSS 19.0 Statistical software analyzes H. pylori infection and eradication failure related influencing factors. According to the analysis, the investigators can provide a scientific basis for local formulation of correct and effective H. pylori prevention and control strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Perform 13-UBT,
2. Be able to understand the content of the questionnaire and answer the questions accurately,
3. Permanent residents of Xi'an area,
4. No previous HP eradication treatment,
5. Agree to join the group and sign the informed consent form,
6. Aged between 18-70.

Exclusion Criteria:

1. Complicated with serious cardiovascular, respiratory, blood, liver, kidney, nerve or endocrine system diseases,
2. Mental disease,
3. Gastric or esophageal surgery history,
4. Severe atypical hyperplasia of gastric epithelium, gastric malignant tumor or other malignant diseases
5. Pregnant or lactating women,
6. Patients with history of penicillin allergy,
7. Allergy to rabeprazole, bismuth dose, clindamycin,
8. Have taken proton pump inhibitors,H2 receptor antagonists, within 2 weeks before participating in the inspection,
9. Have taken herbs that have bacteriostatic effect or antibiotic or bismuth agents within 4 weeks before participating in the inspection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Infection rate | 1 year
  The infection rate is defined as the proportion of patients diagnosed positive among all subjects undergoing 13-UBT.(On the 13-UBT,if the result DOB≥4. 0‰, it can be determined that the subject is H. pylori positive; DOB <4. 0‰,the subject is H. pylori negative)
The Affecting factors of Helicobacter pylori infection is investigated by questionnaire statistics. | 1 year
  The questionnaire refers to "National Helicobacter pylori Research Questionnaire", which is designed by the Department of Epidemiology and Health Statistics, Peking University School of Medicine.And the questionnaire includes general situation, basic situation, living environment and living habits, personal disease history, related symptoms,and family history, etc.Through logistic regression analysis to calculate OR value and P value, to understand the relationship between Helicobacter pylori infection and the factors involved in the questionnaire.
Eradication rate | 1 year
  H. pylori-positive patients are given PPI quadruple therapy,and after 4-6 weeks of completing eradication therapy, 13C-UBT is performed.Eradication rate is defined as the ratio of the number of subjects who become negative after taking the eradication drug to the number of all subjects who take the eradication drug.
The Affecting factors of Helicobacter pylori eradication failure is investigated by questionnaire statistics. | 1 year
  The questionnaire refers to "National Helicobacter pylori Research Questionnaire", which is designed by the Department of Epidemiology and Health Statistics, Peking University School of Medicine.And the questionnaire includes general situation, basic situation, living environment and living habits, personal disease history, related symptoms,and family history, etc.Through logistic regression analysis to calculate OR value and P value, to understand the relationship between Helicobacter pylori eradication failure and the factors involved in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Zhao, MD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The second affiliated hospital of Xi'an Jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No